CLINICAL TRIAL: NCT03298529
Title: Study on Glycemic and Insulin Index Values of Five Types of Pasta With Different Flour Content, and Egg Components
Brief Title: Glycemic Index of Traditional Egg Pasta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Gioacchino Leandro, Head of Gastroenterology, Director of the Service of Clinical Nutrition, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IG2017C
Record Dates: First submitted 2017-09-12; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Glycemic Response; Insulinemic Response; Healthy Subjects
Keywords: Glycemic index; Insulinemic index; Traditional egg pasta
MeSH Terms: interventions — Albumins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Traditional egg pasta (Experimental): Traditional egg pasta. 12 healthy subjects, after a 10 to 12-hour overnight fasting period, will assume "fettuccine" pasta made with 8 eggs/kg flour. The serving size is calculated to contain 50 g of carbohydrates according to nutritional analysis of the product.
  Interventions: Other: glucose solution; Other: Traditional egg pasta
- Pasta with only eight egg whites/kg flour (Experimental): Pasta with only eight egg whites/kg flour. 12 healthy subjects, after a 10 to 12-hour overnight fasting period, will assume "fettuccine" pasta with only eight egg whites/kg flour. The serving size is calculated to contain 50 g of carbohydrates according to nutritional analysis of the product.
  Interventions: Other: glucose solution; Other: Pasta with eight egg whites/kg flour
- Pasta with four eggs/kg flour (Experimental): Pasta with four eggs/kg flour. 12 healthy subjects, after a 10 to 12-hour overnight fasting period, will assume "fettuccine" pasta with four eggs/kg flour. The serving size is calculated to contain 50 g of carbohydrates according to nutritional analysis of the product.
  Interventions: Other: glucose solution; Other: Pasta with four eggs/kg flour
- Hyperproteic pasta (with added gluten and albumin) (Experimental): Hyperproteic pasta (with added gluten and albumin). 12 healthy subjects, after a 10 to 12-hour overnight fasting period, will assume "fettuccine" pasta with added gluten and albumin. The serving size is calculated to contain 50 g of carbohydrates according to nutritional analysis of the product.
  Interventions: Other: glucose solution; Other: Hyperproteic pasta (with added gluten and albumin)
- Pasta with only four egg whites/kg flour (Experimental): Pasta with only four egg whites/kg flour. 12 healthy subjects, after a 10 to 12-hour overnight fasting period, will assume "fettuccine" pasta with only four egg whites/kg flour. The serving size is calculated to contain 50 g of carbohydrates according to nutritional analysis of the product.
  Interventions: Other: glucose solution; Other: Pasta with only four egg whites/kg flour

INTERVENTIONS:
Other: glucose solution — 12 healthy subjects, aged 18-65 years, after a 10 to 12-hour overnight fasting period will assume standard food, a glucose solution at 50%
Other: Traditional egg pasta — 12 healthy subjects, aged 18-65 years, after a 10 to 12-hour overnight fasting period will assume traditional pasta, with 8 eggs/kg flour. The serving size must contain 50 g of carbohydrates, calculated according to nutritional label
  Arms: Traditional egg pasta
Other: Pasta with eight egg whites/kg flour — 12 healthy subjects, aged 18-65 years, after a 10 to 12-hour overnight fasting period will assume pasta, with eight egg whites/kg flour. The serving size must contain 50 g of carbohydrates, calculated according to nutritional label
  Arms: Pasta with only eight egg whites/kg flour
Other: Pasta with four eggs/kg flour — 12 healthy subjects, aged 18-65 years, after a 10 to 12-hour overnight fasting period will assume pasta, with four egg whites/kg flour. The serving size must contain 50 g of carbohydrates, calculated according to nutritional label
  Arms: Pasta with four eggs/kg flour
Other: Hyperproteic pasta (with added gluten and albumin) — 12 healthy subjects, aged 18-65 years, after a 10 to 12-hour overnight fasting period will assume pasta with added gluten and albumin.The serving size must contain 50 g of carbohydrates, calculated according to nutritional label
  Arms: Hyperproteic pasta (with added gluten and albumin)
Other: Pasta with only four egg whites/kg flour — 12 healthy subjects, aged 18-65 years, after a 10 to 12-hour overnight fasting period will assume pasta with four egg whites/kg flour. The serving size must contain 50 g of carbohydrates, calculated according to nutritional label
  Arms: Pasta with only four egg whites/kg flour

SUMMARY:
The glycemic index (GI) compares the plasma glucose response to a specific amount of carbohydrates with the response induced by the same amount of carbohydrates from a standard carbohydrate source, pure glucose in our case. The GI is defined as the incremental area under the curve (iAUC) for blood glucose after consumption of a test food divided by the iAUC of a reference food containing the same amount of carbohydrates. GI is based on the physiologic functions of food carbohydrates rather than on their chemical structure, allowing to a more accurate classification. Several studies found that the regular consumption of low glycemic meals reduces the risk of developing diabetes, insulin-resistance, cardiovascular and neoplastic diseases.

GI was originally developed for insulin-resistant subjects. The maintenance of stable blood glucose levels is a challenge for people with diabetes and pre-diabetes and is also beneficial for the general population, as reported by several studies.

Low-GI diets have been shown to:

* stabilize blood sugar levels
* improve body weight
* better control appetite
* improve memory
* reduce the risk of cardiovascular diseases
* reduce the risk of some forms of cancer According to Walter Willet, nutrition researcher at the Harvard School of Public Health, an excess of sugars and refined starches stimulates insulin hypersecretion, hunger pangs and frequent snacking, slowing down lipid metabolism and making people physically less active.

This project aims to evaluate the glycemic index of five different types of pasta with the same format, named "Fettuccine", but with different composition (the pasta format is related to GI variations). The different types of pasta vary for flour and egg composition. However, having the same format, the GI will change only in response to the percentage content of the ingredients used to produce pasta. In particular, the aim is to measure egg's effect, distinct in yolk and white, on the glycemic and insulin response of healthy subjects.

DETAILED DESCRIPTION:
The five types of pasta to be tested are produced by the so called "La Campofilone" Company (Ficiarà, Campofilone, Marche), a national excellence in the production of traditional egg. Every pasta is designed and realized with the scientific support of two consultants: Prof. Paolo De Cristofaro, endocrinologist, diabetologist and professor at the School of Specialization in Food Science and Nutrition at the University of Chieti, and Prof. Giampiero Sacchetti, biotechnologist at the Marche Polytechnic University. Specifically, the products to be tested are:

1. Traditional Fettuccine, original recipe (8 eggs/kg flour) currently available on the market;
2. Pasta with only 8 egg whites/kg flour;
3. Pasta with 4 eggs/kg flour;
4. Hyperproteic pasta (with added gluten and albumin);
5. Pasta with only 4 egg whites/kg flour.

Each phase of the project will be implemented in accordance with the Jenkins and Wolever protocol (World Health Organization-Food and Agriculture Organization of the United Nations,1998). 12 healthy subjects, aged 18-65 years, will be recruited. After a 10 to 12-hour overnight fasting period, standard food (a glucose solution) and food test (the different types of fettuccine La Campofilone) will be administered to volunteers, organized into groups of two or three people.

Both test food administrations and standard food administrations will take place on a different day. The standard food consists of 50 g of glucose dissolved in oligomineral water, the test food consists of a portion of pasta containing 50 g of available carbohydrates. Blood samples for determination of glycemia and insulinemia will be taken at time 0 and then at 15, 30, 45, 60, 90 and 120 minutes from the beginning of the test or standard food intake. Three glucose response curves will be performed on each subject (this allows to obtain an average value of the subject's response to glucose over time) while a single test with the food to be tested will be done. Blood samples will be analyzed at the Service of Medical Laboratory Analysis of the Hospital "S. De Bellis". Glucose and insulin values will be used to calculate the glycemic and insulin index of each product. For each type of tested pasta, a detailed report will be drawn up, complete with graphs of glycemic response for each subject. Each report will include the glycemic and insulin index of the product under review.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* pregnancy and breast feeding
* athletes
* current pharmacological therapy or pharmacological therapy interrupted less than 3 months before recruitment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
glicemic index | 6 months
  to measure glicemic index of each type of pasta

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda ospedaliera Specializzata in Gastroenterologia Saverio de Bellis, Castellana Grotte, Bari, Italy